CLINICAL TRIAL: NCT03283423
Title: Image-guided Lymphadanectomy in AMIGO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID and OR access
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry); KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Principal Investigator, Ali Tavakkoli, Associate Surgeon, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002535
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Lymphadenopathy Retroperitoneal; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Image Guided Arm (Experimental): Will receive Image guided lymph node biopsy
  Interventions: Device: Image-guided Lymphadanectomy in AMIGO

INTERVENTIONS:
Device: Image-guided Lymphadanectomy in AMIGO — Image guided laparoscopic lymph node biopsy

SUMMARY:
To perform image-guided laparoscopic intra-abdominal lymph node biopsy with goal of minimizing surgical risk and improving accuracy of biopsy.

DETAILED DESCRIPTION:
Only the superficial lymph nodes are accessible to physical examination, and assessment of deeper nodes, such as those in the abdomen, requires radiological imaging. As a result, abdominal CT and PET scanning of patients with a history of malignancy or concerns for a new diagnosis of cancer is an important diagnostic test. As well as looking for distant metastasis, the images are carefully assessed for evidence of intra-abdominal lymphadenopathy, which can be a marker of new or recurrent cancer. If such nodes are identified, they often require a biopsy for further evaluation.

The lymph nodes located in the abdomen or the retroperitoneum are not easily accessible for percutaneous biopsy, often requiring an abdominal exploration which can be done either laparoscopically or via laparotomy. The laparoscopic approach represents a better approach that is associated with reduced surgical risks and complications as well as a quicker recover. In fact in many cases, the laparoscopic approach can be done as a day surgery procedure.

Although non-invasive imaging technologies such as computed tomography (CT) scanning, magnetic resonance imaging (MRI), and positron emission tomography (PET) scanning can be useful in the diagnosis of lymphadenopathy, they often provide an estimate of the location of the nodes, and exact localization of the lymph node of interest can be challenging. The surgeons rely on anatomical landmarks which can be distorted during laparoscopy and to help reduce the rate of false negative lymph node biopsy, the surgeons often perform intra-operative histological assessment of the lymph nodes (Frozen Section) which can be time consuming and in itself associated with diagnostic errors. The uncertainty about the exact location of the node of interest often leads to extensive surgical dissection, biopsy of multiple nodes, and sometimes repeat surgery. During the dissection, care must be taken to avoid injury to the neighboring structures, such as blood vessels, nerves or adjacent organs. In cases, where an intra-operative dissection occurs, or lymph nodes can not be identified, the laparoscopic surgery is converted to open surgery.

Using the unique capabilities of the AMIGO suite, investigators aim to test intra-operative image guidance to help them identify diseased intra-abdominal lymph nodes, allowing for more precise and safer surgeries. The improved accuracy will allow investigators to perform surgeries with minimal dissection and reduced complications while improving biopsy rates and enhancing ability to accurately stage intra-abdominal malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before any trial related procedure is undertaken that is not part of the standard patient management
* Subjects aged ≥ 18 years. Selected patients must have a confirmed or suspected diagnosis of disease in the abdomen or retroperitoneum, with scheduled confirmatory surgical biopsy.
* Subjects must have had a CT, PET examination or MR examination of acceptable quality at Brigham and Women's Hospital within the prior month

Exclusion Criteria:

* Severely impaired renal function with an EGFR < 30 mL/min/body surface area
* Evidence of any significant, uncontrolled comorbid condition that could affect compliance with the protocol or interpretation of the results, which is to be judged at the discretion of the PI
* History of hypersensitivity or other contraindication to contrast media
* Contraindication to general anesthesia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of lymph node biopsy | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ali Tavakkoli, MD, Principal Investigator — Brigham and Women's Hopistal
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No